CLINICAL TRIAL: NCT02976311
Title: Comparison of Inflammatory Reactions Following Two Different Cesarean Surgery Techniques; The Modified Misgav-Ladach Versus the Pfannenstiel-Kerr Technique
Brief Title: Comparison of Inflammatory Responses Subsequent to Different Cesarean Section Techniques
Acronym: C/S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hatice Akkaya, doctor, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E52332816_51
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Delivery; Cesarean Delivery; Inflammation
Keywords: inflammatory reaction; IL-6; TNF; Misgav Ladach technique; Pfannenstiel-Kerr technique; cesarean delivery; cesarean technique
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misgav-Ladach (Active Comparator): cesarean section(C/S) via the modified 'Misgav-Ladach' technique
  Interventions: Procedure: cesarean section(C/S) via the modified Misgav-Ladach technique
- Pfannenstiel-Kerr (Active Comparator): cesarean section(C/S) via the 'Pfannenstiel-Kerr' technique
  Interventions: Procedure: cesarean section via the Pfannenstiel-Kerr technique

INTERVENTIONS:
Procedure: cesarean section(C/S) via the modified Misgav-Ladach technique — the first consecutive 44 patients underwent C/S via the modified Misgav-Ladach technique
  Arms: Misgav-Ladach
Procedure: cesarean section via the Pfannenstiel-Kerr technique — the second consecutive 44 patients underwent C/S via the Pfannenstiel-Kerr technique
  Arms: Pfannenstiel-Kerr

SUMMARY:
In this study, the investigators aimed to find out whether there are any differences in inflammatory reactions occured subsequent to two different cesarean delivery techniques; modified Misgav-Ladach vs Pfannenstiel-Kerr techniques.

DETAILED DESCRIPTION:
Cesarean section is one of the most undertaken operations in women of childbearing age. However, there is not a unique cesarean surgery technique. Pfannenstiel , reported his own technique in 1897. Because of the applicability of the technique, it went down well among obstetricians. After three decades, Kerr evolved this technique, and Pfannenstiel-Kerr technique became the method of choice until late 70's. In 1972, Stark et al defined the Misgav Ladach technique and in the following years this technique became popular among obstetricians. In late 80's Misgav Ladach technique was modified and started to be more popular. But, still Pfannenstiel-Kerr technique continued to be used frequently and studies comparing clinical outcomes of these two techniques were conducted for several times. However, the inflammatory responses which occured subsequent to application of these techniques were not investigated. This is the first study investigating the inflammatory response emerged after different cesarean surgery techniques.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section for the first time
* Term,singleton pregnancy

Exclusion Criteria:

* Any inflammatory disease
* Any pregnancy complication; IUGR,preeclampsia,preterm labor,preterm premature rupture of membranes
* Pregnancies <37weeks gestational age

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
IL-6 | 24 hours
  percentage of difference in serum IL-6 levels just before the beginning of the surgery and at the 24th hour of the surgery
TNF-alpha | 24 hours
  percentage of difference in serum IL-6 levels just before the beginning of the surgery and at the 24th hour of the surgery

IPD SHARING:
Plan to Share IPD: Yes
If needed